CLINICAL TRIAL: NCT00984074
Title: A Pilot Study of Functional Mapping and Brain Perfusion Imaging in Patients Receiving Base of Skull and Brain Radiotherapy: Developing Neurocognitive Functional Organs At Risk for Individualized Conformal Radiotherapy
Brief Title: MRI Mapping in Planning Radiation Therapy to the Base of Skull and Brain in Patients With Nonmetastatic Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000654169; 808258
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer
Keywords: stage III salivary gland cancer; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Tongue Neoplasms | interventions — Diffusion Tensor Imaging; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: blood-oxygen-level-dependent functional magnetic resonance imaging
Procedure: diffusion tensor imaging
Procedure: dynamic contrast-enhanced magnetic resonance imaging
Procedure: functional magnetic resonance imaging
Radiation: intensity-modulated radiation therapy
Radiation: radiation therapy treatment planning/simulation

SUMMARY:
RATIONALE: Diagnostic procedures, such as specialized types of magnetic resonance imaging (MRI), may help in planning radiation therapy that does less damage to normal tissues.

PURPOSE: This phase I trial is studying using functional MRI to see how well it works in planning radiation therapy in patients undergoing radiation therapy to the base of the skull and/or brain for nonmetastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility of applying established MRI techniques to map functional anatomic regions at potential risk in irradiated normal brain tissue of patients undergoing radiotherapy to the base of the skull and brain for head and neck neoplasms.
* To determine changes in cerebral blood flow and blood volume with perfusion MRI techniques in irradiated regions of the brain as a function of the radiation dose.

OUTLINE: Patients undergo MRI perfusion imaging and functional (fMRI) (standard structural imaging sequences, diffusion tensor imaging, arterial spin labeled perfusion imaging at rest, blood oxygen level dependent, and dynamic susceptibility contrast perfusion weighted MRI) at baseline and 3 and 6 months after completion of radiotherapy. Patients may perform tasks for fMRI studies, including finger tapping, photic stimulation with a flashing light, solving math problems, comparing shapes, giving a speech, or listening to and reciting lists of words during fMRI image acquisition. Patients also undergo daily fractionated intensity-modulated radiotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed head and neck cancer that requires radiotherapy to the base of the skull
* No evidence of metastatic disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 1 year
* Not pregnant
* Negative pregnancy test
* Able to undergo standard CT simulation and radiotherapy treatment planning and delivery, including the capacity to comply with standard immobilization devices to the head and neck for daily irradiation
* Able to undergo standard MRI and deemed capable of complying with the immobilization needs and tasks required for functional MRIs
* No claustrophobia
* No patients with pacemakers, metal fragments in the eye, or certain metallic implants

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Base of skull and brain patients
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Feasability, as assessed by the proportion of study patients with functional regions identified within the brain as receiving exit irradiation | 90 days

SECONDARY OUTCOMES:
Summary parameters of the dose volume histograms to the functional regions identified | One year
Cerebral blood flow and blood volume quantitated by relative measures normalized to regions of the brain not receiving any irradiation | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Harry Quon, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials